CLINICAL TRIAL: NCT06753591
Title: Clinical Characteristics and Outcomes of Patients with Premature Acute Myocardial Infarction in Serbia - a Multicenter National Study
Brief Title: PRemature Acute Myocardial Infarction Register of Serbia
Acronym: PRAMIRS
Status: Recruiting | Type: Observational
Sponsor: Cardiology Society of Serbia (Other)
Responsible Party: Sponsor
Other Study IDs: 01/2024
Record Dates: First submitted 2024-12-18; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute Myocardial Infarction; Premature; Young Adults; National Registry
MeSH Terms: conditions — Acute Coronary Syndrome; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Frozen samples for the potential substudies on genetics and non-standard laboratory analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This observational multicentric national study aims to understand better acute myocardial infarction (heart attack) in young adults aged 45 years or younger in Serbia. By analyzing patient characteristics, medical history, test results, and treatment outcomes, the research seeks to identify factors contributing to heart attacks in this population and improve prevention and treatment strategies.

Participants will undergo routine tests during hospitalization, and specific blood samples will be collected for advanced analyses, including genetic testing. Follow-up will include periodic check-ins to monitor health outcomes.

The study will also explore differences in heart attack causes and outcomes in younger individuals compared to older populations, focusing on risk factors like smoking, cholesterol levels, and genetic predisposition.

Participation is voluntary, and all collected data will remain confidential.

DETAILED DESCRIPTION:
Study Overview This national, multicenter study combines retrospective and prospective analyses to investigate AMI in patients aged ≤ 45 years in Serbia. The primary aim is to characterize the clinical, demographic, and angiographic profiles of these patients, identify specific risk factors, and evaluate treatment outcomes. The findings aim to inform prevention, early diagnosis, and treatment strategies for premature AMI.

Objectives

Primary Objectives:

Determine the incidence and prevalence of AMI in this population. Analyze demographic characteristics and the prevalence of standard atherosclerotic risk factors (e.g., smoking, diabetes, hypertension, and socioeconomic status).

Examine angiographic findings, including obstructive or non-obstructive coronary artery disease and other abnormalities.

Secondary Objectives:

Assess atherosclerotic plaque characteristics using OCT or IVUS imaging. Evaluate the prevalence of spontaneous coronary artery dissection (SCAD) and comorbid conditions like chronic kidney disease and autoimmune diseases.

Investigate genetic predispositions (e.g., thrombophilia, familial hypercholesterolemia) and metabolic markers like homocysteine.

Monitor treatment outcomes, including major adverse cardiovascular events (MACE) during hospitalization and at follow-ups.

Design and Methodology

The study adheres to the Universal Definition of Myocardial Infarction and includes detailed data collection:

Demographics: age, gender, socioeconomic status, and rural vs. urban residency. Clinical Data: chest pain characteristics, ECG findings, and laboratory markers like lipids, homocysteine, and inflammatory markers.

Imaging and Diagnostics: echocardiography, angiography, OCT/IVUS imaging, and cardiac MRI for MINOCA cases.

Therapeutics: Analysis of treatment methods, including interventions, antiplatelet agents, and anticoagulants.

Study Population

Inclusion Criteria: Patients aged ≤ 45 years diagnosed with AMI who provide informed consent.

Exclusion Criteria: Patients aged > 45 years. Sample Size and Data Analysis Approximately 200 participants will be enrolled annually, with a target of 1,000 participants over five years. Data will be analyzed using statistical methods to identify predictors of adverse outcomes and evaluate survival rates.

Ethical Considerations This study complies with ethical standards and protects patient rights and data confidentiality. Participation is voluntary, and patients may withdraw at any time without affecting their care.

Significance The study aims to close a critical knowledge gap regarding premature AMI, contributing to improved prevention and management strategies in young adults at the national level.

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≤ 45 years. Clinical and laboratory diagnosis of acute myocardial infarction (AMI) based on the Universal Definition of Myocardial Infarction.

Voluntary participation with signed informed consent.

Exclusion Criteria:

Patients aged > 45 years.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This national, multicentric, retrospective and prospective analysis would include patients with acute myocardial infarction (AMI) aged ≤ 45 years in Serbia
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Incidence and Prevalence of AMI in Patients Aged ≤ 45 Years in Serbia | From 01.January 2021.year to 31.December 2026.
  The incidence and prevalence of AMI among patients aged ≤ 45 years in Serbia will be reported over the study period, expressed as the number of new and existing cases per 100,000 individuals annually Unit of Measure: "Cases per 100,000 individuals per year."
Demographic Characteristics and Prevalence of Atherosclerotic Risk Factors in Young AMI Patients | From 01.January 2021.year to 31.December 2026.
  The demographic distribution (e.g., age, gender, socioeconomic status) and prevalence of standard atherosclerotic risk factors (e.g., smoking, diabetes, hypertension, hyperlipidemia) among AMI patients aged ≤ 45 years will be analyzed.
  Unit of Measure: "Percent of participants with each risk factor."
Angiographic Characteristics in Young AMI Patients | From 01.January 2021.year to 31.December 2026.
  The presence and extent of obstructive and non-obstructive coronary artery disease, coronary lesions, dissection, and vasospasm will be assessed using angiographic findings.
  Unit of Measure: "Percent of participants with each angiographic characteristic."

SECONDARY OUTCOMES:
Characteristics of Atherosclerotic Plaque Using OCT or IVUS | From 01.January 2021.year to 31.December 2026.
  Plaque characteristics, including degree of fibrosis, necrosis, calcification, and vulnerability, will be evaluated in a subset of patients using OCT or IVUS imaging.
  Unit of Measure: "Percent of plaques with specific characteristics (e.g., fibrosis, calcification)."
Prevalence of SCAD in Young AMI Patients | From 01.January 2021.year to 31.December 2026.
  The prevalence of SCAD, including angiographic subtypes defined by current guidelines, will be assessed among participants.
  Unit of Measure: "Percent of participants diagnosed with SCAD."
Prevalence of Comorbidities in Young AMI Patients | From 01.January 2021.year to 31.December 2026.
  The prevalence of comorbid conditions such as kidney disease, chronic lung diseases, systemic autoimmune diseases, and specific chronic therapies will be assessed.
  Unit of Measure: "Percent of participants with each comorbidity."
Prevalence of Inherited or Acquired Thrombophilia in MINOCA Patients | From 01.January 2021.year to 31.December 2026.
  The presence of inherited or acquired thrombophilia in patients with myocardial infarction with non-obstructive coronary arteries (MINOCA) will be analyzed using genetic and laboratory tests.
  Unit of Measure: "Percent of MINOCA participants with thrombophilia."
Prevalence of Familial Hypercholesterolemia in Young AMI Patients | From 01.January 2021.year to 31.December 2026.
  The prevalence of familial hypercholesterolemia in the study population will be determined using genetic testing and clinical diagnostic criteria.
  Unit of Measure: "Percent of participants diagnosed with familial hypercholesterolemia."
Mean Homocysteine Levels in Young AMI Patients | From 01.January 2021.year to 31.December 2026.
  Homocysteine concentrations will be measured in all participants to determine average levels and their correlation with AMI.
  Unit of Measure: "Mean homocysteine concentration (µmol/L)."
Treatment Modalities and Interventions in Young AMI Patients | From 01.January 2021.year to 31.December 2026.
  The number and type of percutaneous coronary interventions (PCI), number of stents implanted, and antiplatelet/anticoagulant therapies will be assessed.
  Unit of Measure: "Percent of participants receiving specific interventions."
Number of Participants Experiencing MACE During Hospitalization, at 1 Month, and 1 Year Post-AMI | From 01.January 2021.year to 31.December 2026.
  The number of participants experiencing MACE, including cardiovascular death, recurrent MI, revascularization, stroke, heart failure, or hospitalization, will be recorded during hospitalization at 1-month and 1-year follow-ups.
  Unit of Measure: "Number of participants experiencing MACE."

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Djokovic, MD, PhD, Principal Investigator — Cardiology Society of Serbia, Belgrade, Serbia; Svetlana Apostolovic, Md, PhD, Principal Investigator — Cardiology Society of Serbia, Belgrade, Serbia
Locations (11):
- Serbia (11):
  - Military Medical Academy 1, Belgrade
  - University Hospital Center Zvezdara, Belgrade
  - University Hospital Center Bezanijska kosa, Belgrade
  - University Hospital Center Zemun, Belgrade
  - Military Medical Academy 2, Belgrade
  - General Hospital Studenica, Kraljevo
  - University Clinical Center Nis, Niš
  - Institute for cardiovascular diseases Vojvodina, Novi Sad
  - General Hospital Prokuplje, Prokuplje
  - General Hospital Vrbas, Vrbas
  - General Hospital Zrenjanin, Zrenjanin

IPD SHARING:
Plan to Share IPD: Yes
For the purposes of meta statistical analysis
Supporting Information: Study Protocol, ICF
Time Frame: From 30.December 2026
Access Criteria: Principal Investigators of other national registries involving AIM in young adults